CLINICAL TRIAL: NCT00986466
Title: Effects of Vitamin D and Exercise in Preventing Falls of Elderly Women
Brief Title: Vitamin D and Exercise in Falls Prevention
Acronym: DEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Academy of Finland (Other); Tampere University Hospital (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Kirsti Uusi-Rasi, Ph.D./ senior researcher, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R09090; SA131524
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Falls Prevention; Prevention of Fall-related Injuries
Keywords: exercise; falls; physical functioning; vitamin D; mobility function; neuromuscular functioning¨; quality of life; number of fallers; fall-related injuries including bone fractures; bone mass
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- exercise with vitamin D 800 IU/d (Experimental)
  Interventions: Dietary Supplement: exercise and vitamin D supplementation
- exercise with placebo (Active Comparator)
  Interventions: Dietary Supplement: exercise and vitamin D supplementation
- no exercise with vitamin D 800 IU/d (Active Comparator)
  Interventions: Dietary Supplement: exercise and vitamin D supplementation
- no exercise with placebo (Placebo Comparator)
  Interventions: Dietary Supplement: exercise and vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: exercise and vitamin D supplementation — 20 µg (800 IU) of vitamin D per day for two years supervised training two times a week for 12 months, and once a week during the next 12 months
  Other Names: Mini-Sun; strength training; balance training; mobility training
  Arms: exercise with vitamin D 800 IU/d
Dietary Supplement: exercise and vitamin D supplementation — placebo per day for two years supervised training two times a week for 12 months, and once a week during the next 12 months
  Other Names: Mini-Sun; strength training; balance training; mobility training
  Arms: exercise with placebo
Dietary Supplement: exercise and vitamin D supplementation — 20 µg (800 IU) of vitamin D per day for two years no supervised training (maintenance of their current level of physical activity)
  Other Names: Mini-Sun; strength training; balance training; mobility training
  Arms: no exercise with vitamin D 800 IU/d
Dietary Supplement: exercise and vitamin D supplementation — placebo per day for two years no supervised training (maintenance of their current level of physical activity)
  Other Names: Mini-Sun; strength training; balance training; mobility training
  Arms: no exercise with placebo

SUMMARY:
The aim of the study is to investigate the effects of exercise and vitamin D supplementation on reducing falls and injuries in community-dwelling, independent-living women aged 70-79 years of age. The investigators will test the following hypothesis:

1. Exercise including strength, balance and mobility training will improve muscle functioning and body balance, and thus reduce falls by 30% compared with non-exercisers.
2. Vitamin D intake will improve muscle functioning and thus prevent falls by 30% compared with placebo.
3. Together vitamin D and exercise have a stronger influence on fall prevention than either used alone.
4. Training improves mobility functions and bone health.
5. Supervised training twice a week with daily home training will improve physical functioning thus resulting in reduced fear of falling.
6. Reduced fear of falling and improved physical functioning help older people to stay physically active, which further improve their quality of life.

DETAILED DESCRIPTION:
Falls account for over 80% of all injury-related admissions to hospital among older people. Although there is evidence that both exercise and vitamin D improve neuromuscular and cognitive function, and may thus reduce the risk of falls and fractures, these two factors have never been evaluated together in a clinical trial. This study is a randomized 24-month intervention in elderly women. The investigators hypothesize that exercise and vitamin D supplementation reduce falls and injuries including fractures in community-dwelling, independent-living women 70-79 years of age. The eligible participants will be randomly assigned into one of four groups:

1. exercise with vitamin D
2. exercise with placebo
3. no exercise with vitamin D
4. no exercise with placebo. The rational of this study is to provide important information on how to maintain and improve physical functioning and thus prevent falls and fractures of elderly people. In addition, if fear of falling can be declined with this program, it will further help elderly people to keep physically active and maintain their functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 70-80 years old
* lives at home independently
* has fallen at least once during the previous year
* no contraindication to exercise
* understands the procedures of the study
* has been informed of X-ray radiation doses of the DXA and pQCT investigations

Exclusion Criteria:

* moderate-to-vigorous exercise more than 2 hours per week
* regular use of vitamin D, or calcium + vitamin D supplements
* a recent fracture (during preceding 12 months)
* contraindication or inability to participate in the exercise program
* marked decline in the basic activities of daily living (ADL-test)
* cognitive impairments (Mini Mental State Examination, MMSE-test < 18)
* persons with chronic disease conditions, such as Parkinson's disease

Ages: 70 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 409 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
number of falls | 24 months

SECONDARY OUTCOMES:
number of fallers | 24 months
bone mass | 24 months
fall-related injuries including bone fractures | 24 months
physical functioning | 24 months
fear of falling | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kirsti Uusi-Rasi, PhD, Principal Investigator — UKK Institute for Health Promotion Research
Locations (2):
- Finland (2):
  - University of Helsinki, Helsinki
  - UKK Institute for Health Promotion Research, Tampere

REFERENCES:
- [Background] Uusi-Rasi K, Kannus P, Karinkanta S, Pasanen M, Patil R, Lamberg-Allardt C, Sievanen H. Study protocol for prevention of falls: a randomized controlled trial of effects of vitamin D and exercise on falls prevention. BMC Geriatr. 2012 Mar 26;12:12. doi: 10.1186/1471-2318-12-12. PMID 22448872
- [Result] Patil R, Uusi-Rasi K, Pasanen M, Kannus P, Karinkanta S, Sievanen H. Sarcopenia and osteopenia among 70-80-year-old home-dwelling Finnish women: prevalence and association with functional performance. Osteoporos Int. 2013 Mar;24(3):787-96. doi: 10.1007/s00198-012-2046-2. Epub 2012 Jun 12. PMID 22688541
- [Result] Uusi-Rasi K, Karinkanta S, Heinonen A, Sievanen H. Improved femoral neck BMD in older Finnish women between 2002 and 2010. Maturitas. 2013 Jul;75(3):241-5. doi: 10.1016/j.maturitas.2013.04.001. Epub 2013 Apr 30. PMID 23642771
- [Result] Patil R, Uusi-Rasi K, Pasanen M, Kannus P, Karinkanta S, Sievanen H. Cross-sectional studies and methodology: reply to comment by Erkoyun. Osteoporos Int. 2013 Feb;24(2):743. doi: 10.1007/s00198-012-2134-3. Epub 2012 Sep 29. No abstract available. PMID 23052929
- [Result] Patil R, Uusi-Rasi K, Pasanen M, Kannus P, Karinkanta S, Sievanen H. Sarcopenia prevalence: reply to comment by Perez-Zepeda et al. Osteoporos Int. 2013 Mar;24(3):799. doi: 10.1007/s00198-012-2092-9. Epub 2012 Aug 1. No abstract available. PMID 22850867
- [Derived] Patil R, Kolu P, Raitanen J, Valvanne J, Kannus P, Karinkanta S, Sievanen H, Uusi-Rasi K. Cost-effectiveness of vitamin D supplementation and exercise in preventing injurious falls among older home-dwelling women: findings from an RCT. Osteoporos Int. 2016 Jan;27(1):193-201. doi: 10.1007/s00198-015-3240-9. Epub 2015 Jul 24. PMID 26205890
- [Derived] Patil R, Uusi-Rasi K, Tokola K, Karinkanta S, Kannus P, Sievanen H. Effects of a Multimodal Exercise Program on Physical Function, Falls, and Injuries in Older Women: A 2-Year Community-Based, Randomized Controlled Trial. J Am Geriatr Soc. 2015 Jul;63(7):1306-13. doi: 10.1111/jgs.13489. Epub 2015 Jun 26. PMID 26115073
- [Derived] Uusi-Rasi K, Patil R, Karinkanta S, Kannus P, Tokola K, Lamberg-Allardt C, Sievanen H. Exercise and vitamin D in fall prevention among older women: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):703-11. doi: 10.1001/jamainternmed.2015.0225. PMID 25799402
- [Derived] Patil R, Uusi-Rasi K, Kannus P, Karinkanta S, Sievanen H. Concern about falling in older women with a history of falls: associations with health, functional ability, physical activity and quality of life. Gerontology. 2014;60(1):22-30. doi: 10.1159/000354335. Epub 2013 Oct 8. PMID 24107382